CLINICAL TRIAL: NCT04214938
Title: Hypertonic Saline Enhances The Field of View of Clinicians and Ease of Procedures: A Double Blind, Randomized, Controlled Trial Comparing the Efficacy of Intranasal Hypertonic Saline, Xylometazoline, Lidocaine, and Isotonic Saline
Brief Title: Hypertonic Saline Enhances The Field of View of Clinicians and Ease of Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merih Onal, Associate Professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 15.01.2015
Record Dates: First submitted 2019-12-23; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Nasopharyngeal Diseases
Keywords: hypertonic saline solutions; lidocaine; oxymetazoline; isotonic saline; discomfort
MeSH Terms: conditions — Nasopharyngeal Diseases | interventions — halofantrine

STUDY DESIGN:
Intervention Model Description: A Double Blind, Randomized, Controlled Trial
Who Masked: Participant, Investigator
Masking Description: The caregiver administering the nasal spray, the subject, and the otolaryngologist carrying out nasendoscopy were all uninformed as to the type of spray employed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hypertonic sea water (Active Comparator): The patient was applied intranasal hypertonic sea water (3.5% sodium chloride) before the nasoendoscopy procedure.
  Interventions: Other: Intranasal solutions application were done including one solution for per patient before nasoendoscopy procedure according to randomization
- Lidocaine (Active Comparator): The patient was applied intranasal Vemcaine as TLA (10% lidocaine; AstraZeneca, Södertälje, Sweden) before the nasoendoscopy procedure.
  Interventions: Other: Intranasal solutions application were done including one solution for per patient before nasoendoscopy procedure according to randomization
- Xylometazoline (Active Comparator): The patient was applied intranasal Otrivine (0.1% xylometazoline hydrochloride, GlaxoSmithKline, Brentford, UK ) before the nasoendoscopy procedure.
  Interventions: Other: Intranasal solutions application were done including one solution for per patient before nasoendoscopy procedure according to randomization
- 0.9% Sodium chloride (Placebo Comparator): The patient was applied intranasal placebo (0.9% sodium chloride) before the nasoendoscopy procedure.
  Interventions: Other: Intranasal solutions application were done including one solution for per patient before nasoendoscopy procedure according to randomization

INTERVENTIONS:
Other: Intranasal solutions application were done including one solution for per patient before nasoendoscopy procedure according to randomization — Hypertonic sea water, Vemcaine, Otrivine, and a placebo were applied by intranasal before the nasoendoscopy procedure for improving the field of view of clinician and reducing the patient discomfort.
  Other Names: intranasal hypertonic sea water (Ancient Secrets, USA); intranasal lidocaine (Vemcaine AstraZeneca, Södertälje, Sweden); intranasal xylometazoline (Otrivine, GlaxoSmithKline, Brentford, UK); intranasal isotonic saline (Deva, Istanbul, TR)

SUMMARY:
Transnasal Flexible Pharyngolaryngoscopy (NPL) is one of the most common and fundamental evaluation procedures in otolaryngologist's practice, performed in both outpatient and ward settings.In the studies the desired properties for an effective topical agent to be used in patients undergoing NPL. To date, only a local anesthetic and/or decongestant substance is applied to the nostrils to relieve pain. However, to date, no studies have been performed in which intranasal hypertonic saline was used prior to nasal endoscopy.

DETAILED DESCRIPTION:
NPL is a technique that has been used for more than 100 years and increases brightness, magnification and the ability to take still and video images (3). NPL is a simple, safe, cost-effective, and generally well-tolerated procedure. However, a portion of patients may refuse to allow the procedure to be repeated as they find it uncomfortable, intolerable, or painful.To date, only a local anesthetic and/or decongestant substance is applied to the nostrils to relieve pain and increase the field of view and to reduce the duration of examination and unpleasant sensations for the patient on NPL procedures.This randomised control trial was undertaken to compare the application of nasal hypertonic sea water (3.5%) with nasal lidocaine 10%, topical nasal decongestant xylometazoline 0.1% (OtrivineTM) and nasal isotonic serum physiologic as placebo group in relation to how they effectively improve the adequacy of the examination and if they reduce pain and discomfort associated with endoscopic nasal examination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who undergone diagnostic nasal endoscopy between 2015- 2017

Exclusion Criteria:

* Had experienced nasal endoscopy before
* Pregnant
* Allergic to either xylometazoline or lidocaine
* Asthma
* Cardiovascular disease
* Rhinitis
* Severe septal deviation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Quality of view, ease of procedure | 2 years
  The primary outcome was to evaluate clinicians' field of the view according to Visual Analog Scale (VAS) questionnaire survey. Shortly after endoscopy, the endoscopist was asked to indicate the degree of quality of view, ease of procedure on a VAS (1: impossible to pass the endoscope, 100: excellent field of view)

SECONDARY OUTCOMES:
Post-op pain | 2 years
  The secondary outcome was to evaluate the patients' pain after the naso-endoscopy procedure according to Visual Analog Scale (VAS) questionnaire survey. Shortly after endoscopy, subjects were asked to indicate their degree of pain on a VAS (1: no pain, 100: unbearable pain).
Post-op discomfort | 2 years
  The secondary outcome was to evaluate the patients' discomfort after the nasoendoscopy procedure according to Visual Analog Scale (VAS) questionnaire survey. Shortly after spraying each bottle, subjects were asked to indicate their degree of discomfort on a visual analogue scale (VAS) (1: no discomfort, 100: utmost discomfort). For each spray, one independent scores were obtained from each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Ozkan Onal, Professor, Principal Investigator — Selcuk University